CLINICAL TRIAL: NCT03381105
Title: From PSA to Stockholm3, a Naturalistic Effectiveness Multipart Research Program: Study Part 1
Brief Title: From PSA to Stockholm3: Study Part 1
Acronym: PSA2STHLM3/1
Status: Active, not recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: SUSID_637
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: Diagnostics, over-diagnosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PSA and Stockholm3 — The new Stockholm3 test and traditional PSA test

SUMMARY:
This part of the project aims to analyze the effectiveness of the Stockholm3 test in regular clinical practice, both in general practice and in the specialist health care, as a tool for detecting patients who need further diagnostics for prostate cancer.

DETAILED DESCRIPTION:
Background:

Prostate cancer constitutes about 15 % of new cases of cancer among men globally, but about 27 % of all new cases of cancer in men in Norway. It is also the leading cause of cancer death among men, and nearly 1100 Norwegian men died from prostate cancer in 2014. However, only about 30 percent of new cases have an aggressive form of the disease. Therefore, the challenge is to detect and distinguish patients with aggressive disease from patients who have a low risk cancer.

The Prostate-Specific Antigen (PSA) is currently the main test used in primary care to detect and prioritize patients for further diagnostics. PSA is used for screening in many countries, but the Norwegian authorities consider the harms of using PSA for screening purposes (over-diagnosis and overtreatment) to outweigh the benefits (potentially reduced mortality). Nevertheless, it has been documented that a substantial amount of opportunistic PSA screening takes place in Norway.

At present, a novel test called the Stockholm3 test has been developed. A large prospective study has shown that the efficacy of the Stockholm3 test is superior to PSA, and both the sensitivity and the specificity are substantially higher for Stockholm3 than for PSA.

Aim The aim of this study is to analyze the effectiveness of the Stockholm3 test in regular clinical practice, including both primary care and specialized health care.

Study Design From September 2017, the urological department at Stavanger University Hospital requires a Stockholm3 answer in referrals of patients for further diagnostics of possible prostate cancer.

Comparable clinical data will be collected for a period before - and from a corresponding period after the Stockholm3 test was taken into use.

An analysis will then be carried out where the results from the period where referrals were based primarily on PSA will be compared with the results for the period in which the Stockholm 3 test was used.

Power calculation Based on results from the original Stockholm3 study and aggregated figures regarding PSA testing, prostate biopsies and MRI of the prostate in Stockholm and Stavanger, a statistical power has been calculated. Based on a two-sided alpha at 0.05 (i.e., 5%) and a 90% power the study need about 8000 participants to reliably answer the main study questions. An interim analysis will be conducted in the inclusion phase. A new power calculation will be performed based on the registered data, and the need of participants will be adjusted if necessary.

ELIGIBILITY:
Inclusion Criteria:

* All men where a physicians in regular clinical work finds that there is an indication to take the test

Exclusion Criteria:

* known prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All men at risk of prostate cancer in the 18 municipalities covered by Stavanger University Hospital
Sampling Method: Probability Sample
Enrollment: 13431 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of prostate cancer with Gleason score ≥ 7 / Gleason score ≤ 6 | 9 to 12 months from september 2017 compared with a corresponding period one year earlier
  The percentage of patients whose prostate biopsies showed a Gleason score ≤ 6 or ≥7 among those referred for diagnostics based on a PSA test or a Stockholm3 test

SECONDARY OUTCOMES:
Rate of prostate biopsies among patients tested with PSA and Stockholm3 | 9 to 12 months from september 2017 compared with a corresponding period one year earlier
  The percentage of patients referred for further diagnosis of potential prostate cancer with biopsy among those who were tested with PSA over a period of time, compared to those tested with Stockholm3 for a corresponding period of time

CONTACTS AND LOCATIONS:
Overall Officials: Svein Kjosavik, MS PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gronberg H, Adolfsson J, Aly M, Nordstrom T, Wiklund P, Brandberg Y, Thompson J, Wiklund F, Lindberg J, Clements M, Egevad L, Eklund M. Prostate cancer screening in men aged 50-69 years (STHLM3): a prospective population-based diagnostic study. Lancet Oncol. 2015 Dec;16(16):1667-76. doi: 10.1016/S1470-2045(15)00361-7. Epub 2015 Nov 10. PMID 26563502